CLINICAL TRIAL: NCT07069062
Title: A Multicenter, Open-label Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Clinical Efficacy of HY0001a for Injection in Patients With Advanced Malignant Solid Tumors
Brief Title: A Phase I/Ⅱ Human Study of HY0001a for Injection in Adult Participants With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to a strategic amendment to the protocol, leading to the creation of separate regional studies.
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY0001-101
Record Dates: First submitted 2025-06-26; First posted 2025-07-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product HY0001a for injection (Experimental): HY0010a for injection should be administered at the recommended dosage
  Interventions: Drug: Test product HY0001a for injection

INTERVENTIONS:
Drug: Test product HY0001a for injection — HY0010a for injection should be administered at the recommended dosage

SUMMARY:
This is a multicenter, open-label, phase I/Ⅱ study to evaluate the safety, efficacy, and pharmacokinetic (PK)/pharmacodynamic(PD) characteristics of HY0001a for injection in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase I/II, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of HY0001a for injection in patients with advanced/metastatic solid tumors. HY0001a for injection is administered via intravenous infusion using an accelerated titration method followed by a conventional 3 + 3 study design to identify the maximum tolerated dose (MTD) and dose-limiting toxicities（DLT）. In addition, the maximum-tolerated dose and recommended Phase II dose for HY0001a for injection will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign an informed consent form, understand the study and be willing and able to follow and complete all trial procedures;
* ≥18 years old and ≤75 years old, gender: male or female;
* Patients have histological or cytological diagnosis with advanced solid tumors, cann't benefit from existing standard treatment options;The solid tumors included in the dose-expansion phase are as follows: Cohort 1: Esophageal cancer (patients who have previously received at least two lines of standard therapy);Cohort 2: Non-small cell lung cancer (patients who have previously received at least two lines of standard therapy);Cohort 3: Other tumors, such as cervical cancer, squamous cell carcinoma of the head and neck, pancreatic cancer, gastric adenocarcinoma, gastroesophageal junction adenocarcinoma, breast cancer, etc. (patients who have failed or are intolerant to standard therapy).
* In the dose-escalation phase, patients must have evaluable tumor lesions; in the dose-expansion phase, patients must have at least one measurable tumor lesion (according to RECIST 1.1 version);
* In the dose-escalation phase, enrollment does not require the expression of CDCP1 (CUB domain containing protein 1). In the dose-expansion phase, enrollment is required to be positive for CDCP1
* Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
* Life expectancy ≥3 months;
* Participant must have adequate main organ function;
* Fertile female patients must have a negative serological pregnancy test within 7 days before the first dosing and be willing to use effective birth control/contraception to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Male patients must agree to have no sperm donation plans and to use effective contraceptive methods during the study period until 6 months after the last dose of the study. Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile.

Exclusion Criteria:

* Having received anti-tumor treatments such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, or immunotherapy within 4 weeks prior to the first administration of the study drug
* Known history of severe allergic reactions, or individuals who have experienced an allergic reaction to any of the excipients in the formulation of HY0001a for injection
* Participants who have previously failed treatment with antibody-drug conjugates (ADCs) that use microtubule inhibitors (Monomethyl auristatin E/Monomethyl auristatin F) as toxins
* Participants who have received other investigational drugs or participated in interventional medical device studies within 4 weeks prior to the first administration of the study drug;
* Participants who have received (attenuated) live vaccines within 4 weeks prior to the first administration of the study drug;
* Participants who have undergone major organ surgery (excluding biopsy) within 4 weeks prior to the first administration of the study drug or have experienced significant trauma, or who require elective major organ surgery (excluding biopsy) during the study period;
* Participants who are currently receiving, or who have received treatment with strong CYP3A4 or P-gp inducers or inhibitors within at least one week or five half-lives (whichever is longer) prior to the first administration of the study drug (limited to the dose-escalation phase).
* Participants with uncontrolled, unstable, or active central nervous system (CNS) metastases detected by computed tomography (CT) or magnetic resonance imaging (MRI) during the screening period and before radiological assessment
* Participants with clinically uncontrollable hypertension (defined in this protocol as having a systolic blood pressure > 150 mmHg and/or a diastolic blood pressure > 100 mmHg despite antihypertensive treatment, and which is considered clinically significant by the investigator);
* Participants who have received allogenic tissue/organ transplants in the past;
* Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);Active or chronic hepatitis B or hepatitis C infection; treponema pallidum antibody positive, and confirmed positive test;
* Presence of ophthalmic diseases or symptoms that are deemed by the investigator as not meeting the eligibility criteria at the screening stage.
* Presence of sensory and/or motor neuropathy of Grade ≥2 during the screening period (according to CTCAE Version 5.0)
* Individuals with any of the following cardiac conditions: a. Left ventricular ejection fraction (LVEF) ≤ 50% (Echocardiography, abbreviated as ECHO); New York Heart Association (NYHA) Class III or IV congestive heart failure; b. Significant arrhythmias requiring treatment, including a QTcF (corrected QT interval) ≥ 480 ms measured by electrocardiogram (ECG) (QTcF = QT/(RR^0.33)); c. History of myocardial infarction, unstable angina, or clinically significant valvular disease within 6 months prior to dosing; other cardiac diseases deemed by the investigator as unsuitable for enrollment.
* Presence of other diseases that severely endanger the safety of the participant or affect the participant's ability to complete the trial, such as active gastrointestinal bleeding, active peptic ulcer, intestinal obstruction, intestinal ileus, renal failure, and uncontrolled diabetes (glycated hemoglobin (HbA1c) > 8% during the screening period)
* Participants with active infections deemed inappropriate for entry into the study by the investigator;
* Participants with uncontrolled third-space effusion requiring clinical intervention;
* Participants with a history of drug abuse or medical, psychological, or social conditions that may interfere with study participation or impair the assessment of study outcomes;
* Participant whose toxicities from previous anti-cancer therapy have not resolved, defined as toxicity (hair loss excluded) that has not resolved to grade ≤1 (CTCAE 5.0 version, peripheral neuropathy, ≤grade 2; exclusion criteria specified);
* Female participants who are breastfeeding or have positive urine or blood pregnancy test results during the screening period; female participants who have a planned pregnancy, sperm donation, or egg donation during the study period or within 6 months after the last study drug administration;
* Known history of hypersensitivity to any of the components of the test formulation.
* Participants who have had other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma of the skin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Part One): Incidence and Nature of Dose-Limiting Toxicity (DLT) | 21 days during the first 3-week cycle
  Dose-Limiting Toxicity (DLT) will be defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose Escalation (Part One): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Dose Expansion (Part Two): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR)

SECONDARY OUTCOMES:
Dose Expansion (Part Two): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Dose Escalation and Expansion: Assessment of HY0001a for injection, HY0001a-TAb, and free monomethyl auristatin E (MMAE, i.e., the toxin) Cmax | Up to 2 years
  Maximum concentration observed (Cmax) observed from the pharmacokinetic profile
Dose Escalation and Expansion: Assessment of HY0001a for injection, HY0001a-TAb, and free MMAE (i.e., the toxin) AUC | Up to 2 years
  Area under the concentration versus time curve calculated using the trapezoidal method
Dose Escalation and Expansion: Assessment of HY0001a for injection, HY0001a-TAb, and free MMAE (i.e., the toxin) T1/2 | Up to 2 years
  The time it takes for half the drug concentration to be eliminated calculated using slope of the terminal line
Dose Escalation (Part One): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed complete response (CR) or a Partial Response (PR) determined by Investigator per the Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1
Dose Escalation and Expansion: Duration Of Response (DOR) assessed by investigator per Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 | Up to 2 years
  Duration Of Response (DOR) is defined as the time from the measurement criteria are first met for complete response (CR) /Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease.
Dose Escalation and Expansion: Disease Control Rate (DCR) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Disease Control Rate is defined as the percentage of participants who have achieved CR or PR or have demonstrated stable disease
Dose Escalation and Expansion: Progression-Free Survival (PFS) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Progression-Free Survival (PFS) is defined as the time from the date of first administration of HY0001a to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Dose Escalation and Expansion: Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from the date of first administration of HY0001a to death due to any cause
Immunogenicity assessment indicator: Anti-drug antibodies (ADA) | Up to 2 years
  Incidence, duration, titer of serum anti-HY0001a ADA

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China